CLINICAL TRIAL: NCT06443346
Title: Prospective Registry of EoSinophilic esOphagitis (PRESO)
Brief Title: Prospective Registry of EoSinophilic esOphagitis
Acronym: PRESO
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Alberto Barchi, Medical Doctor, IRCCS San Raffaele
Other Study IDs: PRESO
Record Dates: First submitted 2024-05-30; First posted 2024-06-05 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Eosinophilic Esophagitis — Eosinophilic Esophagitis patients with a proper diagnosis

SUMMARY:
This is a prospective registry of all the Eosinophilic Esophagitis (EoE) patients referred to the third level referral centre of San Raffaele Scientific Institute

DETAILED DESCRIPTION:
Primary objective of the study is to create a registry of all EoE patients with > 18 years of age referring to the Motility and EoE Unit of San Raffaele Hospital, in order to register clinical, endoscopic and histologic data on the disease, to further design and propose future prospective or retrospective studies to increase disease knowledge and foster collaborations with other centers nationally and internationally

ELIGIBILITY:
Inclusion Criteria:

1. Participant is willing and able to give informed consent for participation in the study.
2. The medical product is the standard of care for the patient or the participant is taking the medicinal product according to clinical practice
3. Being diagnosed with EoE as per guidelines of the disease

Exclusion Criteria:

1. No clear diagnosis of EoE
2. Not willing to provide informed consent to the inclusion in the registry

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: EoE patients with a definite diagnosis according to the recent guidelines: >15 eos HPF as peak eosinophils count in at least 1 esophageal location in presence of symptoms of esophageal disfunction, undergoing various treatment and subsequent follow-up visits and endoscopies
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2034-12-31 (Estimated); Study Completion 2044-12-31 (Estimated)

PRIMARY OUTCOMES:
The prospective collection of histologic, endoscopic and clinical data on EoE patients | 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Furuta GT, Katzka DA. Eosinophilic Esophagitis. N Engl J Med. 2015 Oct 22;373(17):1640-8. doi: 10.1056/NEJMra1502863. PMID 26488694
- [Background] Arias A, Perez-Martinez I, Tenias JM, Lucendo AJ. Systematic review with meta-analysis: the incidence and prevalence of eosinophilic oesophagitis in children and adults in population-based studies. Aliment Pharmacol Ther. 2016 Jan;43(1):3-15. doi: 10.1111/apt.13441. Epub 2015 Oct 28. PMID 26510832
- [Background] Mansoor E, Cooper GS. The 2010-2015 Prevalence of Eosinophilic Esophagitis in the USA: A Population-Based Study. Dig Dis Sci. 2016 Oct;61(10):2928-2934. doi: 10.1007/s10620-016-4204-4. Epub 2016 Jun 1. PMID 27250980
- [Background] Dellon ES, Peery AF, Shaheen NJ, Morgan DR, Hurrell JM, Lash RH, Genta RM. Inverse association of esophageal eosinophilia with Helicobacter pylori based on analysis of a US pathology database. Gastroenterology. 2011 Nov;141(5):1586-92. doi: 10.1053/j.gastro.2011.06.081. Epub 2011 Jul 14. PMID 21762663
- [Background] Kottyan LC, Davis BP, Sherrill JD, Liu K, Rochman M, Kaufman K, Weirauch MT, Vaughn S, Lazaro S, Rupert AM, Kohram M, Stucke EM, Kemme KA, Magnusen A, He H, Dexheimer P, Chehade M, Wood RA, Pesek RD, Vickery BP, Fleischer DM, Lindbad R, Sampson HA, Mukkada VA, Putnam PE, Abonia JP, Martin LJ, Harley JB, Rothenberg ME. Genome-wide association analysis of eosinophilic esophagitis provides insight into the tissue specificity of this allergic disease. Nat Genet. 2014 Aug;46(8):895-900. doi: 10.1038/ng.3033. Epub 2014 Jul 13. PMID 25017104
- [Background] Ma C, Schoepfer AM, Safroneeva E; COREOS Collaborators; COREOS Collaborators. Development of a Core Outcome Set for Therapeutic Studies in Eosinophilic Esophagitis (COREOS): An International Multidisciplinary Consensus. Gastroenterology. 2021 Sep;161(3):748-755. doi: 10.1053/j.gastro.2021.04.080. Epub 2021 May 20. No abstract available. PMID 34022180
- [Background] Hahn JW, Lee K, Shin JI, Cho SH, Turner S, Shin JU, Yeniova AO, Koyanagi A, Jacob L, Smith L, Fond G, Boyer L, Lee SW, Kwon R, Kim S, Shin YH, Rhee SY, Moon JS, Ko JS, Yon DK, Papadopoulos NG. Global Incidence and Prevalence of Eosinophilic Esophagitis, 1976-2022: A Systematic Review and Meta-analysis. Clin Gastroenterol Hepatol. 2023 Dec;21(13):3270-3284.e77. doi: 10.1016/j.cgh.2023.06.005. Epub 2023 Jun 17. PMID 37331411